CLINICAL TRIAL: NCT02810665
Title: Repeatability and Concordance of Visual Acuity Level Measured With ETDRS Numeric Charts, ETDRS Landolt C Charts, and Original ETDRS Letter Visual Acuity Charts in Thai Individuals
Brief Title: Repeatability and Concordance of VA Measured With ETDRS Numeric , Landolt C, and Letter Charts in Thai Individuals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Voraporn Chaikitmongkol, Instructor, Chiang Mai University
Other Study IDs: OPT-2558-03133
Record Dates: First submitted 2016-06-16; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Visual Nonspecific
Keywords: Repeatability; Concordance; Agreement; ETDRS visual acuity chart; numeric; Landolt C; Roman alphabet

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal vision group: Individuals with VA 20/20 to 20/25
  Interventions: Behavioral: Visual acuity measurement by ETDRS chart
- Impaired vision group: Individuals with impaired vision: VA of 20/32 to 20/200 due to either cataract, diabetic macular edema, or age-related macular degeneration
  Interventions: Behavioral: Visual acuity measurement by ETDRS chart

INTERVENTIONS:
Behavioral: Visual acuity measurement by ETDRS chart — All participants must complete VA measurement of the study eye using 3 charts including the original ETDRS alphabet, ETDRS Landolt C, and ETDRS numeric charts for 2 times, at least 30 minutes apart.

SUMMARY:
This is a cross-sectional study to determine the repeatability and concordance of visual acuity level measured with the original ETDRS letter, ETDRS Landolt C, and ETDRS numeric chart in Thai individuals.

DETAILED DESCRIPTION:
The ETDRS visual acuity chart has been used as a standard visual acuity measurement chart in ophthalmic clinical trials due to its proven high repeatability comparing to other visual acuity chart. However, the original ETDRS alphabet chart could not be used in every individual around the world, especially those who are non-english speakers. Landolt C chart has been a recommended chart to test visual acuity in those living in a country where English is not a common language, however, some difficulties including right-left confusion occurred when testing with the Landolt C chart, leading to the unreliable results of visual acuity measurement using the Landolt C chart. Recently, the ETDRS numeric chart was introduced by some medical equipment companies but there is limited information regarding the repeatability and concordance of the new ETDRS numeric chart comparing to the original ETDRS alphabet and Landolt C chart.

Therefore, this study aims to determine the repeatability and concordance of visual acuity level measured with the original ETDRS alphabet, the ETDRS Landolt C, and the ETDRS numeric chart. Results from this study would be able to suggest an appropriate ETDRS chart to be used in clinical studies in Thailand or other countries where English is not the native language.

ELIGIBILITY:
Inclusion Criteria:

* Thai nationality
* More than 18 years of age
* Educational level: at least high school
* Able to read English alphabet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with normal vision (VA of 20/20 to 20/25) and decreased vision (VA of 20/32 to 20/200 due to cataract, diabetic macular edema, or age-related macular degeneration) who gave consent to participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Concordance of VA tested with ETDRS alphabet, Landolt C and numeric visual acuity charts | Day 1

SECONDARY OUTCOMES:
Repeatability of VA tested with ETDRS alphabet, Landolt C and numeric visual acuity charts | Day 1
Differences in testing duration of VA measurement across the 3 ETDRS charts | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Voraporn Chaikitmongkol, Muang Chiang Mai, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ricci F, Cedrone C, Cerulli L. Standardized measurement of visual acuity. Ophthalmic Epidemiol. 1998 Mar;5(1):41-53. doi: 10.1076/opep.5.1.41.1499. PMID 9575537
- [Result] Ferris FL 3rd, Kassoff A, Bresnick GH, Bailey I. New visual acuity charts for clinical research. Am J Ophthalmol. 1982 Jul;94(1):91-6. PMID 7091289
- [Result] Kaiser PK. Prospective evaluation of visual acuity assessment: a comparison of snellen versus ETDRS charts in clinical practice (An AOS Thesis). Trans Am Ophthalmol Soc. 2009 Dec;107:311-24. PMID 20126505
- [Result] Ruamviboonsuk P, Tiensuwan M, Kunawut C, Masayaanon P. Repeatability of an automated Landolt C test, compared with the early treatment of diabetic retinopathy study (ETDRS) chart testing. Am J Ophthalmol. 2003 Oct;136(4):662-9. doi: 10.1016/s0002-9394(03)00394-5. PMID 14516806